CLINICAL TRIAL: NCT03602833
Title: Compound 451238 and Radiotherapy in Soft-tissue Sarcoma
Brief Title: Phase I Study Compound 451238 and Radiotherapy in Soft-tissue Sarcoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR 4640; 2017-001316-11 (EudraCT Number)
Record Dates: First submitted 2018-05-18; First posted 2018-07-27 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-06

CONDITIONS: Soft-tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Compound 451238 (Experimental): To assess the safety and tolerability of combining radiotherapy with compound 451238, treating advanced STS.
  Interventions: Drug: Compound 451238

INTERVENTIONS:
Drug: Compound 451238 — Each patient will receive compound 451238 until disease progression unacceptable toxicities.

SUMMARY:
The objective of this trial is to assess the safety and tolerability of combining compound 451238 and radiotherapy, treating advanced STS.

DETAILED DESCRIPTION:
Overall Study Design

This is a single centre open label, non-randomized, non-placebo phase 1 clinical trial to establish the safety and tolerability compound 451238 in combination with radiotherapy in patients with soft tissue sarcomas (STS). STS patients receiving radiotherapy to a tumour deposit above the diaphragm in the thorax, trunk or extremity, will receive radiotherapy. This study will recruit 12 patients and run as a fixed dose trial. Patients will continue on the treatment regimen unless they progress, suffer unacceptable toxicities, or withdraw from the trial.

Treatment Regimen

A maximum of 12 patients will be recruited. The safety and tolerabilty will be assessed in the first 3+3 patients with expansion to 12 patients as tolerated. A minimum gap of 2 weeks will be left between treatment of the first and second patient (with the combination of RT) to mitigate against multiple patients suffering acute toxicity. Patients will be followed for a minimum of 11 weeks from the initiation of radiotherapy with combined compound 451238 for the purposes of acute toxicity monitoring. Late toxicity monitoring will commence from 11 weeks + one day from initiation of radiotherapy with combined compound 451238 and continue until disease progression or initiation of new anti-cancer therapy.

Safety Follow-up - 30 Days

All patients will be required to attend a safety follow-up visit 30 days after the last dose of compound 451238 or before the initiation of a new anti-cancer treatment, whichever comes first.

Extended Safety Follow-up - 90 Days

Given the potential risk for delayed toxicities, an extended safety follow-up visit must be performed up to 90 days after the last dose of compound 451238 administration. The extended safety follow-up will be performed either via a site visit or via a telephone call with subsequent site visit requested in case any concerns noted during the telephone call. All AEs and SAEs that occur prior to the safety follow-up visit should be reported as described in the trial protocol. After the safety follow-up any unresolved AEs at the patient's last visit should be followed up for as long as medically indicated, but without further recording in the CRF.

Follow-up

Patients who discontinue trial treatment for any reason other than disease progression will move into the follow-up phase and will be assessed every 12 weeks by MRI or radiologic imaging to monitor disease status. Every effort will be made to collect information regarding disease status until the start of new anti-cancer therapy, disease progression, death, withdrawal or end of the study. Information regarding post-study anticancer treatment will be collected if new treatment is initiated.

Survival Follow-up

Once a patient experiences confirmed PD or starts a new anti-cancer therapy, the patient moves into the survival follow-up phase and will be followed up every 12 weeks to determine their disease status. This will be done by reviewing their medical notes and/or contacting the patient and/or General Practitioner directly. Patients will remain on this follow-up until death, withdrawal of consent, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of soft tissue sarcoma with at least 2 metastases not suitable for cure using conventional treatments. At least one lesion must be suitable to receive palliative radiotherapy. The radiation tumour target volume must be between the neck and the diaphragm in the thorax, trunk of an extremity.
* Histological confirmed diagnosis of soft-tissue sarcoma .
* Age ≥ 18 years.
* Life expectancy of > 12 weeks.
* At least one site of accessible disease of pre- and post-treatment core biopsies.
* At least two sites of measurable disease on CT
* ECOG Performance Status of ≤ 1.
* Adequate bone marrow function
* Adequate renal function defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula.
* Adequate liver function.
* Written, voluntary informed consent.
* Patients may have received ≥ 1 or more lines systemic therapies. Women of childbearing potential (WOCBP) and male partners of WOCBP must agree to use 2 highly effective methods of contraception from giving informed consent for a period of 28 days prior to administration of first dose of compound 451238, throughout treatment with compound 451238 and for at least 60 days after treatment. Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative pregnancy test ≤ 72 hours prior to Day 1 of study as defined in section 7.3.7.
* Women of childbearing potential include pre-menopausal women and women within the first 2 years of the onset of menopause. Women of childbearing potential must have a negative pregnancy test ≤ 72 hours prior to Day 1 of study as defined in section 7.3.7. See CTFG Contraception Guidance 15.09.2015.
* Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg or 10 mg equivalent prednisone per day
* Administration of steroids through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) are acceptable.
* Patients with a contraindication to MRI (standard of care imaging for extremity disease only) can be entered into the study and will have CT based RECIST 1.1 assessments.
* In patients who have symptoms, when assessed using CTCAE v.4.0, these are of grade 0 or 1 severity only.

Exclusion Criteria:

* Systemic chemotherapy within 28 days prior to study entry.
* Prior systemic therapy.
* Patients who are curable by conventional multidisciplinary management.
* Patients with known central nervous system metastatic disease are ineligible for enrollment.
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
* Patients who have received radiotherapy ≤ 4 weeks prior to Day 1 of study or who have not recovered adequately from side effects.
* Previous radiotherapy within the treatment area.
* Patients who have active infections requiring therapy.
* Patients with a history of Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C. Positive test for HBV surface antigen and / or confirmatory HCV RNA (if anti-HCV antibody tested positive.
* Patients that have a known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
* Patients who received systemic anti-cancer treatment prior to the first dose of study drug within the following time frames:
* Patients who have received biologic therapy within 4 weeks.
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug
* Patients with active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo or resolved childhood asthma/atopy would be exception to this rule. Patients that require inhaled steroids or local steroid injections would not be excluded from the study. Patients with hypothyroidism not from autoimmune disease that is stable on hormone replacement will not be excluded from the study.
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (eg, intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication). xvi. Active autoimmune disease that might deteriorate. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Current severe acute or chronic colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis.
* Women who are pregnant or nursing/breastfeeding.
* Known hypersensitivity to compound 451238.
* Patients with a history of non-infectious pneumonitis that has required a course of oral or intravenous steroids to assist with recovery, or interstitial lung disease.
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Patients requiring steroid replacement doses above physiological requirements will be considered ineligible for this study: allowed up to 20 mg hydrocortisone (or 5 mg of prednisolone) in the morning and 10 mg hydrocortisone (or 2.5 mg prednisolone) in the evening.
* Patients with the risk factors for bowel obstruction or bowel perforation (examples include but not limited to a history of acute diverticulitis, intra-abdominal abscess, abdominal carcinomatosis).
* Patients who have received a live vaccine within 30 days prior to the first dose of trial treatment.
* Previous malignant disease within the last 5 years with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ.
* Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable. xxviii. Patients on anticoagulation medication.
* Patients who have symptoms, which when assessed using CTCAE v.4.0, are of grade 2 severity or above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-11-05 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Determine the safety and tolerability of compound 451238 in combination with radiation therapy in patients with soft-tissue sarcoma as assessed by CTCAE v4.0 at 11 weeks from the start of radiotherapy. | 2 years
  To assess the safety and tolerability of combining radiotherapy with compound 451238 as evidenced by the rate of occurrence of dose limiting toxicities assessed using CTCAE v4.0.
  .

SECONDARY OUTCOMES:
Evaluate local control (LC) | 3 months
  To measure the local control (LC) at 3 months.
To determine progression free survival (PFS) | 1 Year
  To measure progression free survival (PFS) at 6 months and 1 year.
To determine overall survival (OS) | 1 Year
  To measure overall survival (OS) at 6 months and 1 year.
To determine acute toxicity | 11 weeks
  Measure acute ≥ grade 2 toxicity from initiation of radiotherapy and compound 451238 up to 11 weeks following initiation of combined radiotherapy and compound 451238.
To determine late toxicity | 11 weeks plus one day until disease progression
  Measure late ≥ grade 2 toxicity from 11 weeks plus one day after initiation of combined radiotherapy and compound 451238 up to confirmed disease progression or initiation of new anti-cancer treatment therapy.
To measure progression free survival (PFS) in PD-L1 positive population at 6 months and 1 year. | 1 year
  To evaluate progression free survival (PFS) in a PD-L1 positive population.
To measure overall survival (OS) in PD-L1 positive population at 6 months and 1 year. | 1 year
  To evaluate overall survival (OS) in a PD-L1 positive population.

OTHER OUTCOMES:
To evaluate the extent of abscopal effect on local and distant metastasis when compound 451238 and RT are combined. | 2 years
  To assess for evidence of abscopal response using change in value of selected immunological biomarkers.
Identification of immunological biomarkers that correlate with response to therapy. | 2 years Description: To evaluate whether radiation therapy combined with compound 451238results in a measurable change in anti-tumour immunity.
  To evaluate which immunological biomarkers best predict measurable anti-tumour response to radiation therapy combined with compound 451238.

CONTACTS AND LOCATIONS:
Overall Officials: Shane Zaidi, Principal Investigator — MRCP FRCR
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Summary of Product Characteristics — https://www.medicines.org.uk/emc/product/8453